CLINICAL TRIAL: NCT06329726
Title: Long-Term Behavioral and Cognitive Outcomes of Deep Brain Stimulation in Patients With Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: NeuroPsico_DBS&PD
Record Dates: First submitted 2024-03-06; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Deep Brain Stimulation; Cognitive dysfunction; Mood; Anxiety; Quality of life
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Anxiety Disorders | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD - undergone DBS: Patients with Parkinson's disease treated with DBS of the subthalamic nucleus
  Interventions: Diagnostic Test: Clinical examinations and clinical scales administration
- PD - not undergone DBS: Patients with Parkinson's disease not treated with DBS
  Interventions: Diagnostic Test: Clinical examinations and clinical scales administration

INTERVENTIONS:
Diagnostic Test: Clinical examinations and clinical scales administration — Psychometric assessment of cognitive and behavioral outcomes

SUMMARY:
The goal of this observational study is to evaluate the long-term effect of DBS-STN on cognitive and behavioral outcomes in Parkinson's disease (PD) patients.

PD patients will be assessed over time using tests, questionnaires and standardized clinical scales. An initial assessment (T0) and annual follow-up assessments will be carried out for 5 years.

Researchers will compare data collected from patients with DBS versus patients with best medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients candidates for DBS of the subthalamic nucleus
* Parkinson's disease patients with best medical treatment

Exclusion Criteria:

* patients unable to complete study assessments

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2031-12-15 (Estimated); Study Completion 2032-12-15 (Estimated)

PRIMARY OUTCOMES:
Long-term characterization of DBS-STN on cognitive outcomes | Annual assessments up to 5 years
  Cognitive impairment change from baseline until 5 years in Montreal Cognitive Assessment (MoCA; min. 0, max. 30, higher score means better outcome) [Time Frame: Annual assessments up to 5 years]
Beck Depression Inventory | Annual assessments up to 5 years
  Depressive symptoms change from baseline to 5 year (BDI-II, min 0, max 63, higher score means worse outcome)
State-Trait Anxiety Inventory | Annual assessments up to 5 years
  Anxiety symptoms change from baseline to 5 year (STAI, min 20, max 80, higher score means worse outcome)
Questionnaire for Impulsive-Compulsive Disorders in Parkinson | Annual assessments up to 5 years
  Impulsivity change from baseline to 5 years (QUIP, min 0, max 112, higher score means worse outcome)
Pittsburgh Sleep Quality Index | Annual assessments up to 5 years
  Sleep Quality change (PSQI, min 0, max 21, higher score means poorer sleep quality)
Parkinson's Disease Questionnaire-8 | Annual assessments up to 5 years
  Quality of life change from baseline to 5 years (PDQ-8, min 0, max 100, higher score means worse outcome)
Minnesota Multiphasic Personality Inventory 2-RF | Annual assessments up to 5 years
  Personality change from baseline to 5 years (MMPI-2-RF, cut-off: T>65 for clinical scales)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Mameli, Dr, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy, Italy